CLINICAL TRIAL: NCT04593459
Title: Probiotic Dietary Intervention in Polycystic Ovary Syndrome (PCOS) - A Randomized Controlled Trial
Brief Title: Probiotic Intervention in PCOS
Acronym: ProPCO-RCT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of Graz (Other)
Collaborators: Institut AllergoSan (Unknown); Winclove Probiotics B.V. (Industry)
Responsible Party: Principal Investigator, Barbara Obermayer-Pietsch, Professor, MD, Medical University of Graz
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 160120200001; 2020-000228-20 (EudraCT Number)
Record Dates: First submitted 2020-10-12; First posted 2020-10-20 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2024-03

CONDITIONS: Polycystic Ovary Syndrome
Keywords: PCOS; Probiotic; Metformin; RCT
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — Probiotics; Metformin

STUDY DESIGN:
Intervention Model Description: Probiotic vs placebo (double-blinded) vs metformin (open-label)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Only the probiotic and placebo are blinded, metformin is an open intervention arm
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Probiotic (Experimental): Probiotic product consisting of these 7 bacterial strains:
  * Lactobacillus salivarius W57
  * Lactobacillus casei W56
  * Lactobacillus rhamnosus W71
  * Lactococcus lactis W58
  * Enterococcus faecium W54
  * Lactobacillus plantarum W62
  * Lactobacillus acidophilus W22
  Additional ingredients: Corn starch, maltodextrin, fructo-oligosaccharides, galacto-oligosaccharides, polydextrose, plant proteins, potassium chloride, magnesium sulfate, bacterial strains, manganese sulfate, lactose, 2000 IU vitamin D
  Participants ingest one sachet of powder (5 grams) in 200 ml of water per day for 6 months
  Interventions: Dietary Supplement: Probiotic
- Placebo (Placebo Comparator): Similar to probiotic product in optics and smell, less ingredients and no bacterial strains or vitamin D
  Ingredients: Corn starch, maltodextrin, potassium chloride, magnesium sulphate, manganese sulphate
  Interventions: Dietary Supplement: Probiotic Placebo
- Metformin (Active Comparator): Metformin is an established drug for treating PCOS-related symptoms. The investigators are comparing the probiotic not only to a placebo group, but also to the benchmark treatment.
  Participants in the metformin arm will start treatment with 500 mg daily for the first week, then increasing the dose to 2x500 mg daily for the duration of the intervention.
  Interventions: Drug: Metformin Hydrochloride

INTERVENTIONS:
Dietary Supplement: Probiotic — See Arm description
  Arms: Probiotic
Drug: Metformin Hydrochloride — See Arm description
  Arms: Metformin
Dietary Supplement: Probiotic Placebo — See Arm description
  Arms: Placebo

SUMMARY:
The investigators are conducting a double-blinded randomized controlled trial to determine whether a probiotic mixture is effective in reducing PCOS-related symptoms. For this purpose, 180 participants will be recruited in three intervention arms (Probiotic, Placebo and Metformin), with 60 participants per arm. The intervention period will last 6 months, with extensive medical history, blood work, urine and stool analysis at the beginning and the conclusion of the trial.

ELIGIBILITY:
Inclusion Criteria:

* Polycystic Ovary Syndrome diagnosed based on at least two out of three rotterdam criteria: hyperandrogenism, polycystic ovarian morphology, oligo-/anovulation
* signed informed consent

Exclusion Criteria:

* Missing or withdrawn consent
* Hyperandrogenism of a cause other than PCOS (Cushing´s syndrome, hyperprolactinemia, adrenal tumours, congenital adrenal hyperplasia, rare genetic disorders)
* Pregnancy or nursing period (first 6 months after giving birth)
* Soy or other allergies with respect to study procedures
* Diabetes mellitus type 1
* Chronic inflammatory bowel disease, history of cancer in the gastrointestinal tract or acute gastrointestinal infection
* Any malignancies that required treatment within the last 3 years prior to study procedures
* Any other chronic disease requiring medical check-ups or hospital treatments at least once every three months (exception: diabetes mellitus type 2)
* Major surgery in the gastrointestinal tract (e.g. colectomy, gut segment excision with stoma surgery, Whipple´s surgery.) Surgical removal of the appendix and/or the gall bladder is NOT considered major surgery.
* Therapy with antidiabetic drugs (metformin, sulfonylureas, dipeptidyl peptidase 4 (DPP-4) inhibitors, Glucagon-like peptide 1 (GLP-1) analogs, sodium-glucose-cotransporter 2 (SGLT-2) inhibitors, insulin variants) within the last six months prior to study procedures
* Therapy with proton pump inhibitors within the last six months prior to study procedures
* Therapy with hormonal contraceptives or systemic (oral) intake of steroids within the last six months prior to study procedures
* Oral or intravenous therapy with antibiotics less than three months before the onset of study procedures
* Alcohol and/or drug abuse

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 112 (Actual)
Dates: Start 2020-11-03 (Actual); Primary Completion 2023-10-16 (Actual); Study Completion 2023-10-16 (Actual)

PRIMARY OUTCOMES:
Free testosterone | 6 months
  Changes in free testosterone levels [pg/ml] in serum after intervention

SECONDARY OUTCOMES:
Anti-Müllerian hormone (AMH) | 6 months
  Changes in AMH levels in serum after intervention [ng/ml]
Androstenedione | 6 months
  Changes in androstenedione levels in serum after intervention [ng/ml]
Dehydroepiandrosterone-sulphate (DHEA-S) | 6 months
  Changes in DHEA-S levels in serum after intervention [µg/ml]
17-Hydroxyprogesterone (17-OH-progesterone) | 6 months
  Changes in 17-OH-progesterone levels in serum after intervention [ng/ml]
17-OH-estradiol | 6 months
  Changes in 17-OH-estradiol levels in serum after intervention [ng/ml]
Total testosterone | 6 months
  Changes in total testosterone levels in serum after intervention [ng/ml]
25-OH-cholecalciferol | 6 months
  Changes in 25-OH-cholecalciferol levels in serum after intervention [ng/ml]
Luteinizing hormone (LH), Follicle-stimulating hormone (FSH) | 6 months
  Changes in LH and FSH levels in serum after intervention [mU/ml]
LH to FSH ratio | 6 months
  Changes in LH to FSH ratio after intervention [1]
Insulin | 6 months
  Changes in insulin levels in serum as measured with a two-hour oral glucose tolerance test (75 mg glucose in 300 ml water, blood draws at 0 minutes, 30 min, 60 min and 120 min) [mU/l]
Glucose | 6 months
  Changes in glucose levels in sodium-fluoride plasma as measured with a two-hour oral glucose tolerance test (75 mg glucose in 300 ml water, blood draws at 0 minutes, 30 min, 60 min and 120 min) [mg/dl]
Homeostasis Model Assessment for Insulin Resistance (HOMA-IR) index | 6 months
  Changes in HOMA-IR index (fasting insulin [mU/l] * fasting glucose [mg/dl]/405) after intervention
Glucose mean | 6 months
  Changes in mean glucose levels (measured with oral glucose tolerance test with the formula g=(glucose0 + 2*glucose30 + 3*glucose60 + 2*glucose120)/8 [mg/dl]
Insulin mean | 6 months
  Changes in mean insulin levels (measured with oral glucose tolerance test with the formula i=(insulin0 + 2*insulin30 + 3*insulin0 + 2*insulin120)/8 [mU/l]
Matsuda index | 6 months
  Changes in matsuda index after intervention measured with the formula M=10000/squareroot(glucose0 * insulin0 * glucose mean (see outcome 14) * insulin mean (see outcome 15))
Hirsutism | 6 months
  measured by modified Ferriman-Gallwey-score (mFG-score), ranging from 0 to 36, with 0 being the best possible value and 36 the worst
Body-mass-index (BMI) | 6 months
  BMI measured with the formula BMI=weight [kg]/height² [m]
waist-to-hip ratio | 6 months
  Calculated with the formula: waist circumference/hip circumference [1]
Sucrose-lactulose-mannitol test | 6 months
  Functional gut permeability test consisting of ingesting 20 g sucrose, 5 g mannitol and 10 g lactulose in 100 ml water solution. Measurement of those three component concentrations in urine collected for 5 hours after solution ingestion by the participants. Lactulose to mannitol ratio may be calculated.
Diaminooxidase | 6 months
  Changes in serum diaminooxidase levels after intervention
Stool and serum zonulin | 6 months
  Changes in stool and serum zonulin levels after intervention [ng/ml]
Lipopolysaccharide | 6 months
  Changes in lipopolysaccharide levels after intervention
Soluble cluster of differentiation (sCD14) | 6 months
  Changes in sCD14 levels in serum after intervention
Calprotectin | 6 months
  Changes in stool calprotectin levels after intervention
Bacterial DNA | 6 months
  Changes in bacterial DNA amounts in serum after intervention
Gut lumen and mucosa microbiome composition and metagenomic profile | 6 months
  Measured from stool samples via 16S-RNA gene sequencing
Phytoestrogen production | 6 months
  Changes in daidzein and equol concentrations after intervention [ng/ml] measured in urine samples of participants after ingestion of soy milk
Equol producer status | 6 months
  Equol producer status as determined by the decadic logarithm of the equol/daidzein ratio [1]: A value above -0.5 is defined as an equol producer
Quality of life (QOL) | 6 months
  QOL assessed by General Depression Scale (German: Allgemeine Depressionsskala), German equivalent of the Depression Scale by the Center for Epidemiological Studies (CES-D). The scale ranges from 0 to 60, with 0 being the best possible score and 60 the worst.
QOL | 6 months
  QOL assessed by Beck´s Depression Inventory (BDI), a scale ranging from 0 to 63, with 0 being the best possible score and 63 the worst.
QOL | 6 months
  Quality of Life measured by a PCOS questionnaire ranging from 0 to 156, with 0 being the best possible score and 156 the worst

OTHER OUTCOMES:
Lipid metabolism | 6 months
  Low-density lipoproteins (LDL), high-density lipoproteins (HDL), lipoprotein a (LP(a)), triacylglycerols
Fluorescence-activated cell sorting (FACS) analysis | 6 months
  B cell subtypes measured via FACS from whole blood

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Obermayer-Pietsch, Prof. MD, Principal Investigator — Medical University of Graz, Division of Endocrinology and Diabetology
Locations (1):
- Medical University of Graz, Division of Endocrinology and Diabetology, Graz, Styria, Austria

IPD SHARING:
Plan to Share IPD: Yes
For research and cooperation purposes, pseudonymized individual participant data may be shared with other researchers, the decision to do so lies with the principal investigator. In case of publication of our results in a peer-reviewed journal, all relevant data will be made publicly accessible without any personal information
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: to be determined
Access Criteria: to be determined

REFERENCES:
- [Background] Lindheim L, Bashir M, Munzker J, Trummer C, Zachhuber V, Leber B, Horvath A, Pieber TR, Gorkiewicz G, Stadlbauer V, Obermayer-Pietsch B. Alterations in Gut Microbiome Composition and Barrier Function Are Associated with Reproductive and Metabolic Defects in Women with Polycystic Ovary Syndrome (PCOS): A Pilot Study. PLoS One. 2017 Jan 3;12(1):e0168390. doi: 10.1371/journal.pone.0168390. eCollection 2017. PMID 28045919
- [Background] Haudum C, Lindheim L, Ascani A, Trummer C, Horvath A, Munzker J, Obermayer-Pietsch B. Impact of Short-Term Isoflavone Intervention in Polycystic Ovary Syndrome (PCOS) Patients on Microbiota Composition and Metagenomics. Nutrients. 2020 Jun 1;12(6):1622. doi: 10.3390/nu12061622. PMID 32492805
- [Derived] Borzan V, Riedl R, Obermayer-Pietsch B. Probiotic vs. placebo and metformin: probiotic dietary intervention in polycystic ovary syndrome - A randomized controlled trial. BMC Endocr Disord. 2023 Apr 17;23(1):82. doi: 10.1186/s12902-023-01294-6. PMID 37062834